CLINICAL TRIAL: NCT02130583
Title: Skills to Enhance Positive Affect in Suicidal Adolescents
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Shirley Yen, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH101272 (NIH)
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Affect Skills Training (Experimental): Individual sessions (3-4) delivered on the inpatient unit, focused on psycho-education regarding positive affect and mood monitoring and teaching of skills to attend to positive affect such as mindfulness, gratitude, and savoring. In-person sessions are followed by weekly phone calls and daily text messages for one month, with option to extend.
  Interventions: Behavioral: Positive Affect Skills Training
- Treatment as Usual (Active Comparator): Participants will follow the intervention plan laid out in their discharge summary, but do not receive any individual sessions regarding positive affect. Upon discharge, they will receive generic text messages regarding healthy habits for one month, with option to extend.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Positive Affect Skills Training — Individual sessions (3-4) delivered on the inpatient unit, focused on psycho-education regarding positive affect and mood monitoring and teaching of skills to attend to positive affect such as mindfulness, gratitude, and savoring. In-person sessions are followed by weekly phone calls and daily text messages for one month, with option to extend.
  Arms: Positive Affect Skills Training
Behavioral: Treatment as Usual — Participants will follow the intervention plan laid out in their discharge summary, but do not receive any individual sessions regarding positive affect. Upon discharge, they will receive generic text messages regarding healthy habits for one month, with option to extend.
  Arms: Treatment as Usual

SUMMARY:
The prevalence of suicidal behaviors in adolescents remains unacceptably high and is a significant public health concern. The investigators propose a new treatment approach in which skills to increase positive emotions are taught to the most vulnerable at-risk adolescents, those admitted to an inpatient psychiatric unit due to suicide risk. The investigators believe that teaching skills to increase positive emotions will lead to better problem-solving, increased social support, and other benefits which will serve as protective factors and decrease suicide risk.

DETAILED DESCRIPTION:
The prevalence of suicidal behaviors in adolescents remains unacceptably high. Reviews of published randomized controlled trials (RCTs) for adolescent suicidality conclude that treatments to date have been minimally efficacious. The preponderance of interventions focus on crisis intervention, underlying psychiatric disorders, regulating negative affect and reducing cognitive distortions. However, our pilot work and other recent data suggest the importance of considering how low positive affectivity contributes to suicide risk independent of other risk factors and may be another mechanism that leads to suicidal behaviors. Our model is based on Fredrickson's empirically-supported Broaden and Build model which asserts that the function of positive affect (PA) includes helping individuals thrive by improving social supports, problem-solving, and personal resilience. Each of these areas is instrumental in decreasing suicidal behavior. We propose that PA increases survival directly by decreasing suicidal ideation and indirectly by increasing social support and problem-solving. In this R34 treatment development grant we seek to develop a novel, individual skills-based, PA intervention, delivered adjunctively to treatment as usual (TAU), targeting the highest risk adolescents - those hospitalized due to suicide risk. We focus on three strategies that have been demonstrated to increase sustainable (vs. transient) PA in community and depressed adults: meditation, gratitude, and savoring. There are several ways to practice each strategy; we take into account patient preferences in a personalized approach in which patients select the practice(s) that fits best with their needs and circumstances. We propose using multiple means of intervention delivery that includes text messaging, to reinforce in-vivo practice. Our intervention, Skills To Enhance Positivity Program (STEP) includes two phases: a) in-person phase consisting of 3 individual in-person sessions and 1 joint parent session during the inpatient hospital stay to teach positive affect skills and develop a personalized intervention; b) remote delivery phase which consists of weekly telephone booster calls and daily text messages over 4 weeks post-discharge. The phone calls will be used to review or adjust personalized intervention components and reinforce use of skills. The text messages will include self-scripted reminders to practice skills and links to online resources. STEP will be tested in an open trial with 20 participants, and after further revision, in a pilot RCT, compared to TAU in a sample of 50 adolescents. The primary goal of this intervention is for patients to increase positive affect by incorporating skills and practices into their normal home-based routines, which we believe will lead to increases in problem-solving and social support and decreases in suicidal ideation. This is a novel intervention for a high-risk acute population via a different mechanism (i.e. PA), and conceptually distinct from other empirically examined theoretical approaches.

ELIGIBILITY:
Inclusion Criteria:

* current hospital admission due to concern of suicide risk
* ability of patient to speak, read, and understand English sufficiently well to complete the procedures of the study
* living at home

Exclusion Criteria:

* active psychotic disorder
* cognitive deficits that preclude full understanding of study materials
* adolescents who have become wards of the state and do not intend to return to the home of their biological or adoptive parents

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09-02 (Actual); Study Completion 2016-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Yen, Ph.D., Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data available upon completion of study by request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 9/1/17
Access Criteria: Please contact PI at 401-444-1915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in this study were adolescents who were hospitalized at a psychiatric hospital in Rhode Island due to concern of suicide risk. The last participant completed the study procedures in September 2016.
Period: Overall Study
Arm/Group | Positive Affect Skills Training | Treatment as Usual
Started | 26 | 26
Completed | 17 | 19
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Affect Skills Training | Treatment as Usual | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.69 (1.1715) | 15.58 (1.206) | 15.63 (1.469)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-identified gender
  Participants
    Female | 15 | 17 | 32
    Male | 10 | 9 | 19
    Other | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Biological Sex
  Participants
    Female | 18 | 18 | 36
    Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dot Probe Task
Description: Dot probe tasks are administered to assess for attentional biases. The task is a computer task in which participants are presented with stimuli (e.g., words) of different valences (positive/negative/neutral) at the same time (e.g., smiling face and a neutral face), followed by a probe (*) on one side. Participants are asked to hit a key that corresponds to the correct side in which the probe appeared. The reaction time of their response is indicative of their attention to the valenced image/word. Trials are counterbalanced so that valences appear equally on each side. Faster reaction time (less milliseconds) to positive images/words indicates an attentional bias for positive stimuli. The scores reported here represent bias scores. Positive scores indicate a bias to positive stimuli, negative scores indicate a bias towards neutral stimuli.
Time Frame: Baseline, 1 month Post Treatment, 4 month Follow-Up
Population: Numbers may differ due to participant attrition and invalid profiles.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- STEP: Study Intervention: Skills to Enhance Positivity
- ETAU: Enhanced Treatment as Usual: Healthy Habits Text Messages
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 26 | 26
milliseconds
  Baseline: number analyzed (Participants) | 26 | 25
  Baseline | 1.56 (18.12) | -1.65 (17.43)
  Post-Treatment: number analyzed (Participants) | 20 | 22
  Post-Treatment | -1.48 (13.85) | 1.23 (18.75)
  Follow-up: number analyzed (Participants) | 16 | 20
  Follow-up | 6.88 (34.12) | -19.8 (40.36)
Statistical Analysis 1: Comparison: STEP vs ETAU; Test type: Superiority; p = .034, ANOVA; Mean Difference (Net) = 2.06

2. Primary Outcome: Modified Differential Emotions Scale (Positive Emotions Sub-scale)
Description: The Modified Differential Emotions Scale is a self-report measure comprised of ratings for positive and negative affect. For example, participants are asked to rate the extent to which they feel "Content, serene, peaceful right now" on a likert scale ranging from 1 (not at all) to 5 (extremely). The scores reported are averages for the positive emotions, and thus can be interpreted as ranging from 1 (not at all) to 5 (extremely). We expected an increase in positive affect ratings following the intervention.
Time Frame: Base, 1 month Post-Treatment, 4 month Follow-Up
Population: Some participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 26 | 26
units on a scale
  Baseline | 1.97 (0.71) | 2.09 (0.71)
  Post-Treatment: number analyzed (Participants) | 21 | 24
  Post-Treatment | 1.95 (0.62) | 2.26 (0.97)
  Follow-up: number analyzed (Participants) | 21 | 21
  Follow-up | 1.98 (0.82) | 2.06 (0.87)

3. Primary Outcome: Suicide Events
Description: Number of participants who have attempted suicide or have had emergency intervention to intercede a suicide attempt.
Time Frame: 1 month, 6 month
Population: Some participants were lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 26 | 26
Participants
  Post-Treatment: number analyzed (Participants) | 21 | 24
  Post-Treatment | 2 | 7
  6 Month Follow Up: number analyzed (Participants) | 17 | 12
  6 Month Follow Up | 5 | 10

4. Secondary Outcome: Suicide Ideation Questionnaire (SIQ)
Description: The Suicidal Ideation Questionnaire is a 30 item self-report measure that was administered to the adolescent to ascertain the frequency of thoughts of death and suicide. Respondents are asked how often they have had these thoughts (e.g., "I thought about killing myself") in the past month ranging from "almost every day" = 1 to "I never had this thought" =7. Scores are then reversed and transformed such that higher scores indicate higher suicidal ideation, with a range of 180 (highest suicidal ideation) to 0 (no suicidal ideation).
Time Frame: Baseline, 1 month Post-Treatment, 4 month Follow-Up
Population: Some participants were lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 26 | 26
units on a scale
  Baseline | 100.04 (44.42) | 106.00 (40.28)
  Post-Treatment: number analyzed (Participants) | 21 | 24
  Post-Treatment | 51.71 (55.24) | 70.96 (42.72)
  Follow-up: number analyzed (Participants) | 21 | 21
  Follow-up | 47.81 (52.96) | 43.24 (45.66)

5. Secondary Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory is a 21 item self-report form of depression but can be and has been administered to the parent to respond about their child. This questionnaire consists of 21 groups of statements. For example, for "Sadness", respondents are asked to select between 0 ("My child does not feel sad."), 1 ("My child feels sad much of the time"), 2 ("My child is sad all the time"), and 3 ("My child is so sad or unhappy that he/she can't stand it."). Higher scores indicate higher depression with a maximum score of 63 and a minimum score of 0.
Time Frame: Baseline, 1 month Post-Treatment, 4 month Follow-Up
Population: Some participants' parents did not participate (e.g. if teen was = 18 y/o); Also, some parents were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 24 | 23
units on a scale
  Baseline: number analyzed (Participants) | 24 | 22
  Baseline | 27.88 (25.79) | 29.77 (8.18)
  Post-treatment: number analyzed (Participants) | 21 | 23
  Post-treatment | 11.56 (11.35) | 20.70 (11.73)
  Follow-Up: number analyzed (Participants) | 17 | 18
  Follow-Up | 11.88 (10.90) | 16.83 (12.66)

6. Secondary Outcome: Columbia Impairment Scale Parent Version
Description: The Columbia Impairment Scale (parent version) is a 13-item scale in which parents are asked to respond about their child's impairment in a variety of domains on a scale of 0 (no problem at all) to 4 (very bad problem). Scores are summed such that higher scored indicate higher functional impairment, with a maximum score of 52 and a minimum score of 0.
Time Frame: Base, 1 month Post-Treatment, 4 month Follow-Up
Population: Some participants' parents did not participate (e.g. if teen was = 18 y/o); Also, some parents were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 24 | 23
units on a scale
  Baseline: number analyzed (Participants) | 24 | 22
  Baseline | 25.79 (10.14) | 26.68 (9.17)
  Post-treatment: number analyzed (Participants) | 21 | 23
  Post-treatment | 17.33 (10.21) | 21.43 (10.59)
  Follow-Up: number analyzed (Participants) | 17 | 18
  Follow-Up | 13.82 (7.23) | 19.78 (8.91)

7. Other Pre Specified Outcome: Hopelessness Scale for Children
Description: The Hopelessness Scale for Children is a 17 item self-report scale with statements (e.g., I want to grow up because I think things will be better) that are rated as either True or False. Some statements are reverse coded. Higher scores indicate higher hopelessness, with a maximum score of 17 and a minimum score of 0.
Time Frame: Baseline, 1 month Post-Treatment, 4 month Follow-Up
Population: Some participants were lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STEP | ETAU
Number analyzed (Participants) | 26 | 26
units on a scale
  Baseline | 7.35 (5.26) | 7.77 (5.00)
  Post-Treatment: number analyzed (Participants) | 21 | 24
  Post-Treatment | 9.24 (5.96) | 10.58 (4.67)
  Follow-up: number analyzed (Participants) | 21 | 21
  Follow-up | 9.71 (5.98) | 11.67 (5.69)

ADVERSE EVENTS:
Time Frame: 1 month, 3 month, 6 months
Arm/Group | Positive Affect Skills Training | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 5/26 | 12/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Affect Skills Training (N=26) | Treatment as Usual (N=26)
Hospitalized for suicidal thoughts and/or behaviors (Psychiatric disorders) | 5 (6) | 9 (13)
Hospitalized for aggressive/assaultive behaviors (Psychiatric disorders) | 0 (0) | 2 (2)
Ran away from home (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study is not powered to observe between group differences or to examine mediators (e.g., increased social support or resources, improved problem-solving). Based on the encouraging preliminary data we are planning a larger trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No